CLINICAL TRIAL: NCT02617732
Title: Effects of Tianqi Capsule on Glucose Variability in Patients With Type 2 Diabetes.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PUMCH-TCM-TQGV-01
Record Dates: First submitted 2015-11-21; First posted 2015-12-01 (Estimated); Last update posted 2015-12-01 (Estimated); Status verified 2015-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: glucose variability; continuous glucose mornitoring system; traditional Chinese medicine
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tianqi capsule (Experimental): a Chinese patent medicine extracted form more than10 kinds of herbs, which was approved to treat type 2 diabetes by CDFA in 2002.
  Interventions: Drug: Tianqi capsule
- placebo (Placebo Comparator): a capsule looks the same as Tianqi capsule, containing starch and other edible compositions.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Tianqi capsule — The patients with type 2 diabetes are divided into two groups, one is experimental group, and the other is placebo group.
  The experimental group patients are treated with Tianqi capsule by oral, 5 pills three times a day
  Other Names: Tianqi Jiangtang Jiaonang, Z20063799
  Arms: Tianqi capsule
Drug: placebo — The patients with type 2 diabetes are divided into two groups, one is experimental group, the other is placebo group.
  The placebo group patients are treated with placebo by oral, 5 pills three times a day
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate the effects and safety of Tianqi Capsule on glucose variability in patients with type 2 diabetes by continuous blood glucose monitoring system.

DETAILED DESCRIPTION:
Diabetes has become a threat to human health and an independent risk factor to macrovascular and microvascular diseases. Large prospective clinical studies have shown a strong relationship between time-averaged mean levels of glycemia as measured by HbA1c and diabetes complications. However, in recent years several pieces of evidence indicated that glucose variability may also contribute to the development of diabetes complications. Thus, glucose variability may become a new target in treatment of diabetes. Traditional Chinese medicine，a kind of multitargeted compound, may contribute to maintaining blood glucose homeostasis in diabetes.

Tianqi capsule(Chinese herbs extract) is a Chinese patent medicine approved to treat T2DM in China. Previous clinical studies have shown that Tianqi capsule could lower blood glucose measured by HbA1c. What's more, Tianqi capsule has also been proved to improve the glycometabolism and lipid metabolism in T2DM and IGT.

This research adopts a randomized, open, parallel double blind, placebo controlled clinical method. The patients, meeting eligibility criteria, are divided into experimental group and placebo group and treated for 12 weeks . A main outcome，glucose variability is detected by continuous blood glucose monitoring system which could obtain continuous and comprehensive blood glucose by "glucose sensor". The influence of Tianqi capsule on glucose variability in type 2 diabetes will be evaluated.

ELIGIBILITY:
Inclusion Criteria

* 18.5kg/m2≤BMI≤35.0 kg/m2;
* meet type 2 diabetes mellitus diagnostic criteria published by 1999 WHO;
* with blood variability, defined as standard deviation of blood glucose more than 3.5mmol／L within 2 days by self-monitoring of blood glucose（SMBG）(more than 5 times per day)
* diabetic duration more than 1 year; in stable condition for more than 4 weeks with unchanged lifestyle and other drugs intervention; （permit taking metformin or sulphonylureas which dosage is unchanged during study period ）
* HbA1c≤10％;
* signed the informed consent form.

Exclusion Criteria:

* have acute diabetes complications （e.g. diabetic ketoacidosis，diabetic hyperosmolar coma,diabetic lactic acidosis,Hypoglycemic coma）
* have severe chronic diabetes complications(e.g. diabetic retinopathy stage 4~6,severe diabetic nephropathy needs dialysis and so on）
* have gastrointestinal disease which have serious influence on digestive function and disorder of absorption
* have other endocrine disease (hyperthyroidism,acromegaly,Cushing's syndrome and so on.)
* have severe heart disease(such as acute myocardium infarction, unstable angina,heart failure NYHA functional classification III or IV）
* have moderate or severe liver function abnormality(ALT,TBil or AST> double upper limit )
* have moderate and severe renal function abnormality(eGFR < 50ml／min)
* blood leukocyte <4.0×10^9/L; blood thrombocyte<90×10^9/L
* taking drugs affecting glucose metabolism,such as glucocorticoid
* have other serious illness which considered to exacerbate and be life-threaten during fellow up period;
* have evidence of mental disorders;
* alcoholics and drug abuse
* females who were pregnant, lactating, planning for pregnancy, or sexually active but with no contraceptive measures;
* have participated in clinical trials within 3 months before;
* other conditions researchers thought to unable to evaluate the curative effect and finish the study.
* allergic to the ingredients of herbs contained in Tianqi capsule

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in mean amplitude of glycemic excursions (MAGE) and mean of daily differences (MODD) at 12 weeks. | 12 weeks
  Glucose variability is evaluated by continuous glucose monitoring system, the main parameters include mean amplitude of glycemic excursions (MAGE)(mmol/L) and mean of daily differences (MODD)(mmol/L). The amplitude of glycemic excursions（AGE）is obtained by continuous glucose, MAGE is calculated using the criterion that both segments of the amplitude of glycemic excursions (AGE) exceed 1 SD, the calculations were carried out as described below, using the formula: MAGE (mg/dL)=∑AGE/n (n=number of glycemic excursions>1 SD). The MODD was calculated as the mean of the absolute difference of glucose values from corresponding times of day from two consecutive days.

SECONDARY OUTCOMES:
Change from baseline in serum lipid and lipoprotein at 12 weeks. | 12 weeks
  Serum lipid and lipoprotein including: triglyceride (TC) (mmol/L); total cholesterol (TG) (mmol/L); low density lipoprotein cholesterol (LDL-C) (mmol/L); high density lipoprotein cholesterol (HDL-C) (mmol/L)
Change from baseline in hemoglobin A1c(HbA1c) at 12 weeks | 12 weeks
Liver Function Examination | 4 weeks
  Liver function examination including alanine aminotransferase (ALT) (U/L) and aspartate transaminase (AST) (U/L).
Renal Function Examination | 4 weeks
  Renal function examination including blood urea nitrogen(BUN)（mmol/L）and urine creatinine(UCr) (mmol/d).

CONTACTS AND LOCATIONS:
Overall Officials: Xiaochun Liang, Doctor, Study Director — Peking Union Medical College Hospital traditional Chinese medicine department
Locations (1):
- Peking Union Medical College Hospital traditional Chinese medicine department, Beijing, Beijing Municipality, China